CLINICAL TRIAL: NCT02132598
Title: A Single-Arm Phase II Clinical Trial of Cabozantinib (XL184) in Patients With Previously Treated Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases With and Without C Met Amplification
Brief Title: Trial of Cabozantinib (XL184) in Non-Small Cell Lung Cancer With Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial stopped due to slow patient accrual.
Sponsor: Liza Villaruz, MD (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Liza Villaruz, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-182
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Metastases to the Brain
Keywords: Lung Cancer; Non Small Cell; Brain metastases; c-MET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Brain Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabozantinib (XL184) (Experimental): Patients will receive cabozantinib at 60 mg orally once daily and continue on treatment until disease progression, death or unacceptable adverse events.
  Treatment cycles are 4 weeks in duration
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib
  Other Names: Cometriq; EXEL-7184; EXEL-02977184; CAS Registry# 1140909-48-3

SUMMARY:
This is an open-label phase II clinical trial designed to allow a preliminary assessment of the efficacy and safety of cabozantinib in unselected Non-Small Cell Lung Cancer (NSCLC) patients with metastases to the brain and in the subset of patients with c-MET amplified Non-Small Cell Lung Cancer with metastases to the brain. Previously treated patients with non-squamous NSCLC who have had brain metastases at any point in their treatment history are eligible for enrollment on this clinical trial. Patients with clinically asymptomatic untreated brain metastases will be allowed on trial at the discretion of the treating investigator. Patients who have undergone treatment for their brain metastases with Whole-Brain Radiation Therapy (WBRT), stereotactic radiosurgery (SRS) or surgery must be clinically stable and recovered from all procedures at the time of study enrollment.

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, open-label study of cabozantinib in subjects with molecularly unselected Non-Small Cell Lung Cancer (NSCLC) with metastases to the brain and in patients with c-MET amplified Non-Small Cell Lung Cancer (NSCLC) with metastases to the brain.

Patients will receive cabozantinib at 60 mg orally once daily and continue on treatment until disease progression, death or unacceptable adverse events. Treatment cycles are 4 weeks in duration.

The primary endpoint is Overall Response Rate (ORR) in both the unselected NSCLC population and the molecularly selected patients on the basis of c-MET amplification.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated patients with non-squamous NSCLC who have had brain metastases at any point in their treatment history are eligible for enrollment on this clinical trial. (Patients must have received at least one regimen for systemic disease which may be cytotoxic or oral tyrosine kinase inhibitor therapy.)

   * Patients with clinically asymptomatic untreated brain metastases will be allowed on trial at the discretion of the treating physician
   * Patients who have undergone treatment for their brain metastases with whole brain radiotherapy, stereotactic radiosurgery, or surgical resection must be clinically stable and recovered from all procedures at the time of study enrollment.
2. Patients must have tumor tissue available for submission that is sufficient to complete c-MET Fluorescence in Situ Hybridization (FISH) studies as well as routine molecular profiling at the UPMC. Patients must agree to submission of these specimens as defined in Section 9.

   * c-MET amplification will be determined by FISH ratio (c-MET/CEP7) > 2.0, based on testing of the primary tumor and/or site of metastatic disease
   * Patients' tumors must undergo testing for Epidermal Growth Factor Receptor (EGFR) exon 19 deletion, EGFR exon 21 L858R substitution, and anaplastic lymphoma kinase (ALK) rearrangements. If positive, patients must have been treated with an appropriate tyrosine kinase inhibitors (TKI) prior to enrolling to the study.
3. The subject has had an assessment of all extracranial disease sites (e.g., by computerized tomography (CT) scan, positron emission tomography-CT, and bone scan as appropriate) within 28 days before the first dose of cabozantinib.
4. The subject must have a baseline brain MRI scan or CT scan of the head (in patients unable to obtain an MRI) within 14 days prior to first dose of cabozantinib.

   * Patients receiving glucocorticoids must be on a stable dose of glucocorticoids during the 5 days prior to the baseline brain imaging.
5. Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
6. Subjects having undergone recent resection or biopsy of an intracranial tumor will be eligible as long as all of the following conditions apply:

   * First dose of cabozantinib occurs at least 28 days after surgery, and the subject has recovered from the effects of surgery
7. Age ≥18 years
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%)
9. Patients must have normal organ and marrow function as defined below: (within 4 days of beginning treatment unless noted otherwise)

   * Hemoglobin ≥9 g/dL
   * Absolute Neutrophil Count (ANC) ≥1,500/mm3 (no CSF support)
   * Platelets ≥100,000/mm3
   * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Bilirubin (Gilbert's Disease) < 3.0 mg/dL
   * Aspartate Aminotransferase (AST) (SGOT) ≤3.0 × ULN
   * Alanine Aminotransferase (ALT) (SGPT) ≤3.0 × ULN
   * Serum creatinine ≤ 1.5 x ULN
   * Creatinine clearance (CrCl) ≥40 mL/min
   * For creatinine clearance estimation, the Cockcroft and Gault equation should be used:
   * Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72)
   * Female: Multiply above result by 0.85 ≤ 1.5 x ULN
   * Lipase (no radiologic or clinical evidence of pancreatitis) < 2.0 x ULN
   * Urine protein/creatinine ratio (UPCR) ≤1
   * Serum phosphorus, calcium, magnesium and potassium ≥ LLN
10. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
11. Women of childbearing potential must have a negative serum pregnancy test at screening.
12. The effects of cabozantinib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 4 months after the last dose of study drug, even if oral contraceptives are used.

Exclusion Criteria:

1. The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies; including investigational biologic agents) within 3 weeks, or nitrosoureas/ mitomycin C within 6 weeks before the first dose of study treatment.
2. The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment.
3. Prior treatment with cabozantinib or other c-MET directed therapy.
4. The subject has received radiation therapy as follows:

   * To the thoracic cavity, abdomen or pelvis within 3 months of the first dose of study treatment or has with ongoing complications or is without complete recovery and healing from prior radiation therapy
   * To bone or brain metastasis within 14 days of the first dose of study treatment
   * To any other site(s) within 28 days of the first dose of study treatment
5. The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment.
6. The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. The subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs.
7. The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment.
8. The subject is receiving concomitant treatment with warfarin, warfarin-related agents, or low molecular weight heparin (LMWH) at the time of study entry at therapeutic doses. Low-dose warfarin (≤ 1 mg/day) or LMWH at prophylactic doses are permitted.
9. The subject has received enzyme-inducing anti-epileptic agents within 2 weeks before the first dose of cabozantinib (e.g., carbamazepine, phenytoin, phenobarbital, primidone). Other enzyme inducing agents prohibited within 2 weeks before the first dose of cabozantinib include rifampin, rifabutin, rifapentin, and St. John's Wort.
10. The subject has experienced any of the following:

    * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment b.Hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment
    * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
11. The subject has radiographic evidence of cavitating pulmonary lesion(s)
12. The subject has tumor abutting, invading or encasing any major blood vessels.
13. The subject has evidence of tumor invading the Gastro Intestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
14. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    * Cardiovascular disorders including:

      * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
      * Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
      * Any history of congenital long QT syndrome
      * Any of the following within 6 months before the first dose of study treatment:

1.unstable angina pectoris 2.clinically-significant cardiac arrhythmias 3.stroke (including Transient Ischemic Attack (TIA), or other ischemic event) 4.myocardial infarction (MI) 5.thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)

* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:
* Any of the following within 28 days before the first dose of study treatment

  1. Intra-abdominal tumor/metastases invading GI mucosa
  2. Active peptic ulcer disease,
  3. Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
  4. Malabsorption syndrome
* Any of the following within 6 months before the first dose of study treatment:

  1. Abdominal fistula
  2. Gastrointestinal perforation
  3. Bowel obstruction or gastric outlet obstruction
  4. Intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment.
* Other disorders associated with a high risk of fistula formation including Percutaneous Endoscopic Gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy.
* Other clinically significant disorders such as:

  * Serious active infection requiring systemic treatment within 28 days before the first dose of study treatment.
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment.
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment.
* History of surgery as follows:

  1. Subjects having undergone recent resection or biopsy of an intracranial tumor will be eligible as long as all of the following conditions apply: First dose of cabozantinib occurs at least 28 days after surgery, and the subject has recovered from the effects of surgery.
  2. Other minor surgery within 28 days of the first dose of cabozantinib if there were no wound healing complications. If there is evidence of wound dehiscence, subjects will be eligible for trial after a minimum of 3 months after surgery to the first dose of cabozantinib, provided complete wound healing is confirmed at least 28 days before the first dose of cabozantinib.
  3. Other major surgery within 2 months of the first dose of cabozantinib if there were no wound healing complications. If there is evidence of wound dehiscence, subjects will be eligible for trial after a minimum of 6 months after surgery to the first dose of cabozantinib, provided complete wound healing in confirmed at least 28 days before the first dose of cabozantinib.
  4. The subject is unable to swallow tablets.
  5. The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before randomization. Note: if initial QTcF is found to be > 500 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.
  6. The subject is pregnant or breastfeeding.
  7. The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
  8. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
  9. The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment. Note: Subjects with a history of early stage or locally advanced non-metastatic prostate cancer within 2 years of the start of study treatment may be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12; Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Villaruz, MD, Principal Investigator — UPCI Department Hematology-Oncology
Locations (1):
- University of Pittsburgh Cancer Institute- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabozantinib (XL184): Cabozantinib - 60 mg orally, once daily (4 weeks treatment cycles)
  Treatment until disease progression, death or unacceptable adverse events.
Period: Overall Study
Arm/Group | Cabozantinib (XL184)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [51.0 to 76.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
c-MET amplification [Count of Participants; unit: Participants] — c-Met, also called tyrosine-protein kinase Met or hepatocyte growth factor receptor (HGFR), is a protein that in humans is encoded by the MET gene. Over-expression of c-Met protein has been associated with poor prognosis in some solid tumors.
  Participants
    Negative | 3
    Positive | 2
Histology [Count of Participants; unit: Participants]
  ADENOCARCINOMA IN SITU, NOS | 1
  ADENOCARCINOMA, NOS | 2
  NON-SMALL CELL CA | 2
Stage of Disease [Count of Participants; unit: Participants] — Stage 0. Cancer in situ; the cancer is only located in the place of origin.
  Stage I. Small tumor with no deep growth into surrounding tissues; no spread to the lymph nodes or other body parts.
  Stage II and Stage III. Larger cancers or tumors that have grown more deeply into surrounding tissue and may have spread to lymph nodes (only).
  Stage IV. Cancer has spread to other body organs (metastasis).
  Participants
    Stage IV | 5
    Stage l-III | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: The proportion of response-evaluable patients who achieve Complete Response (CR) or Partial Response (PR) as best response by RECIST v1.1 criteria. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 12 months
Population: Patients evaluable for response: Received at least one dose of study drug, and, underwent at least one radiologic scan follow-up.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 4
proportion of participants | 0.25 [0.006 to .806]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Proportion of response-evaluable patients that experienced Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) as best response (RECIST v1.1 criteria) per the total study population criteria. Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Stable Disease (SD) is defined as, neither sufficient shrinkage (compared to baseline) to qualify for partial or complete response (CR or PR) nor sufficient increase (taking as reference the smallest sum of diameters at baseline or while on study, whichever is smallest) to qualify for progressive disease (PD).
Time Frame: Up to 16 weeks
Population: As no patients who received at least one dose of study drug and underwent at least one follow-up radiologic scan were able to be evaluated later than 15 weeks, this endpoint cannot be assessed.
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is the time measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression), whichever occurs first, with progression defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 12 months
Population: Only one patient was assessed as having disease progression.
Measure: Number; unit: days
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 1
days | 45

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that patients remain alive, until death from any cause.
Time Frame: Up to 24 months
Population: "All patients" includes all 5 of the patients for whom survival data were available, regardless of c-MET status. "c-MET positive patients" (only) does not include patients for who c-MET status was not positive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 5
months
  All patients | 4.07 [3.09 to NA] — Upper bound of 95% CI not reached
  c-MET positive patients (only): number analyzed (Participants) | 2
  c-MET positive patients (only) | 2.25 [0.43 to NA] — Upper bound of 95% CI not reached

5. Secondary Outcome: Time to Progression (TTP)
Description: Time from initiation of study treatment to disease progression per RECIST v1.1, excluding death from causes unrelated to the disease. As defined by RECIST v 1.1. Progressive disease (PD) is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Until disease progression; Up to 2 years
Population: Only one participant experienced disease progression.
Measure: Number; unit: days
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 1
days | 45

6. Secondary Outcome: Worst Grade of Adverse Events Reported
Description: Worst Grade of Adverse Events Reported as assessed by the investigator. Severity/grade defined by the Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Subjects monitored continuously for Adverse Events (AE's) throughout the study and for 30 days after the last dose of study treatment.
Time Frame: From baseline up to 20 weeks
Population: Patients that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 5
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 4
  Grade 4 | 0
  Grade 5 | 1

7. Secondary Outcome: Worst Grade of AE at Least Possibly Related to Treatment Reported
Description: as for outcome 6
Time Frame: From baseline up to 20 weeks
Population: Patients that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 5
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 5
  Grade 4 | 0
  Grade 5 | 0

8. Secondary Outcome: Worst Grade of AE at Least Probably Related to Treatment Reported
Description: as for outcome 6
Time Frame: From baseline up to 20 weeks
Population: Patients that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 4
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 4
  Grade 4 | 0
  Grade 5 | 0

9. Secondary Outcome: Worst Grade of AE Definitely Related to Treatment Reported:
Description: as for outcome 6
Time Frame: From baseline up to 20 weeks
Population: Patients that received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 1
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after discontinuation of treatment.
Description: Serious Adverse Events are defined as grade 3 and higher toxicity events, per CTCAE v4.0
Arm/Group | Cabozantinib (XL184)
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=5)
Fatigue (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
GGT increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=5)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Pain (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 3
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Serum amylase increased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Ischemia cerebrovascular (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT02132598/Prot_SAP_000.pdf